CLINICAL TRIAL: NCT04782271
Title: Safety, Tolerability and Pharmacokinetic Profile of Different Doses of SYL1801 Ophthalmic Solution in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetic Profile of SYL1801 Eye Drops
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SYL1801_I
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Safety, Tolerability and Pharmacokinetic Profile in Healthy Volunteers; Choroidal Neovascularization
Keywords: Oligonucleotide; siRNA (Small Interfering Ribonucleic Acid); Eye Drops; wet AMD (Age-related Macular Degeneration)
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Interventional, observer-masked, parallel groups, time-lagged trial to study safety, tolerability and PK of SYL1801 sodium in healthy volunteers.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Single administration Low Dose once daily (Experimental): 1 treatment day
  Interventions: Drug: SYL18001 sodium Low dose q.d
- Single administration Middle Dose once daily (Experimental): 1 treatment day
  Interventions: Drug: SYL18001 sodium Middle dose q.d
- Single administration High Dose once daily (Experimental): 1 treatment day
  Interventions: Drug: SYL18001 sodium High dose q.d
- Single administration High Dose twice daily (Experimental): 1 treatment day
  Interventions: Drug: SYL18001 sodium High dose b.i.d
- Multiple administrations Low Dose once daily (Experimental): 7 treatment days
  Interventions: Drug: SYL18001 sodium Low dose q.d
- Multiple administrations Middle Dose once daily (Experimental): 7 treatment days
  Interventions: Drug: SYL18001 sodium Middle dose q.d
- Multiple administrations High Dose once daily (Experimental): 7 treatment days
  Interventions: Drug: SYL18001 sodium High dose q.d
- Multiple administrations High Dose twice daily (Experimental): 7 treatment days
  Interventions: Drug: SYL18001 sodium High dose b.i.d

INTERVENTIONS:
Drug: SYL18001 sodium Low dose q.d — 1 drop in the randomized eye once daily
  Arms: Multiple administrations Low Dose once daily; Single administration Low Dose once daily
Drug: SYL18001 sodium Middle dose q.d — 1 drop in the randomized eye once daily
  Arms: Multiple administrations Middle Dose once daily; Single administration Middle Dose once daily
Drug: SYL18001 sodium High dose q.d — 1 drop in the randomized eye once daily
  Arms: Multiple administrations High Dose once daily; Single administration High Dose once daily
Drug: SYL18001 sodium High dose b.i.d — 1 drop in the randomized eye twice daily
  Arms: Multiple administrations High Dose twice daily; Single administration High Dose twice daily

SUMMARY:
Study of the safety, tolerability and pharmacokinetic profile of different doses of SYL1801 eye drops in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) between 19.5 and 29.0 kg/m2
* Intraocular pressure (IOP) <=21 mmHg
* Best Corrected Visual Acuity (BCVA) >= 70 ETDRS
* Normal corneal and conjunctival assessment
* Normal funduscopy

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test. Females of childbearing potential who will not use a medically acceptable contraceptive method
* Current relevant diseases according to the investigator's judgement.
* Previous relevant chronic processes according to the investigator's judgement
* Relevant visual alterations according to the investigator's judgement
* Administration of systemic medications
* Case history of hypersensitivity to medicinal products or any other allergic process
* Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Ocular tolerability at the site of administration (cornea and conjunctiva) after last instillation of the assigned dose level (1 day of treatment). | 72 hours after last instillation
  Slit lamp evaluation
Ocular tolerability at the site of administration (cornea and conjunctiva) after last instillation of the assigned dose level (7 days of treatment). | 72 hours after last instillation
  Slit lamp evaluation
Determination of the maximum Plasma Concentration [Cmax] | - 15 - 30 minutes, 1- 4 and 24 hours after last administration
Determination of the Area Under the Curve of plasma concentrations until the last extraction time [AUT 0-t] | - 15 - 30 minutes, 1- 4 and 24 hours after last administration

CONTACTS AND LOCATIONS:
Locations (1):
- Sylentis Clinical Trial Site, Madrid, Spain